CLINICAL TRIAL: NCT05383066
Title: Follow-up Registration Management of Anti-angiogenesis Combined With PD-1/PD-L1 Therapy in Patients With Advanced Liver Cancer
Brief Title: Anti-angiogenesis Combined With PD-1/PD-L1 Therapy in Patients With Advanced Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021keyan055
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- those with anti-angiogenesis combined with PD-1/PD-L1 therapy: This study includes patients with advanced liver cancer who can benefit from anti-angiogenesis combined PD-1/PD-L1 treatment and observes the relationship between overall survival and their therpay.

SUMMARY:
To observe and explore the effect of anti-angiogenesis combined with PD-1/PD-L1 therapy in the real world on the survival prognosis of patients with advanced liver cancer, and to summarize the treatment experience of a wide range of people.

DETAILED DESCRIPTION:
This project is a non-interventional, prospective, multicenter, case follow-up registry management, aiming to observe and explore the effect of anti-angiogenesis combined with PD-1/PD-L1 therapy in the real world on the survival prognosis of patients with advanced liver cancer, and to summarize the treatment experience of a wide range of people. Therefore, the data collected and reported in this project will reflect the actual efficacy and safety of anti-angiogenesis combined with PD-1/PD-L1 therapy in patients with advanced liver cancer. 490 patients are planned for follow-up, and enrollment is expected for this program to last for 2 years, starting in December 2021 and ending with the last patient enrollment in December 2023. The treatment period was 24 months, and the patient follow-up was 24 months after the last patient was enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old, male or female;
2. Patients diagnosed with advanced liver cancer, including barcelona stage B, C or Chinese liver cancer guidelines stage IIa, IIb, IIIa, IIIb liver cancer patients;
3. doctors evaluate patients who can benefit from anti-angiogenesis targeted therapy;
4. patients voluntarily join the program and sign informed consent.

Exclusion criteria:

The above selection criteria are not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project is a non-interventional, prospective, multicenter, case follow-up registration management, aiming to observe and explore the impact of real-world anti-angiogenesis targeted therapy on the survival prognosis of patients with advanced liver cancer, and summarize the treatment experience of a wide range of people. Therefore, the data collected and reported in this project will reflect the actual efficacy and safety of anti-angiogenesis targeted therapy in patients with advanced liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 3-4 weeks
  Progression-free survival (PFS) is defined as the time from random assignment in a clinical trial to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 3-4 weeks
  Overall survival was defined as the duration from the date of diagnosis to death or last follow-up, with no restriction on the cause of death.
Objective Response Rate | 3-4 weeks
  Complete response (CR) + partial response (PR) refers to the use of THE RECIST version 1.1 standard to assess the objective efficacy of tumors, including cases of CR and PR.
disease control rate | 3-4 weeks
  Complete response (CR) + partial response (PR) + stable (SD), which refers to the percentage of patients with cr, PR, and SD (≥4 weeks) among patients with measurable efficacy.